CLINICAL TRIAL: NCT05422534
Title: Role of Mitochondrial Dysfunction in the Response to Exercise in Patients With Advance Kidney Disease
Brief Title: CoQ10 and Exercise for Mitochondrial Dysfunction in Advance Kidney Disease
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: University of California, Davis (Other)
Responsible Party: Principal Investigator, Jorge Gamboa, PI, Vanderbilt University Medical Center
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 221073
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: End Stage Renal Disease
Keywords: mitochondrial dysfunction; CoQ10; sarcopenia; frailty; High-intensity interval training (HIIT); exercise; magnetic resonance spectroscopy (P-MRS); physical performance tests
MeSH Terms: conditions — Kidney Failure, Chronic; Mitochondrial Diseases; Sarcopenia; Frailty; Motor Activity | interventions — coenzyme Q10; Ubiquinone; Exercise; Watchful Waiting

STUDY DESIGN:
Intervention Model Description: Randomized, doubled-blinded, 2x2 factorial design, placebo-controlled clinical trial
Who Masked: Participant, Investigator
Masking Description: The randomization will be accomplished through a 2-step procedure. In Step 1, subjects will be randomized to one of the two treatment arms (HIIT and observation) using a permuted-block randomization algorithm. In Step 2, subjects will be randomized to receive either CoQ10 supplement or placebo. Investigators cannot be blinded to HIIT or observation assignments. To avoid bias, study personnel will be blinded to this assignment as much as possible while collecting data at rest during the study visits. Study personnel will be blinded to the study drug assignment that has been determined by the Step 2 randomization schedule.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Observational + placebo (Placebo Comparator): Participants will receive placebo with standard of care or regular activity for 12 weeks.
  Interventions: Drug: Placebo; Behavioral: Observational
- Observational+ CoQ10 (Active Comparator): Participants will receive CoQ10 1800 mg/day with standard of care or regular activity for 12 weeks.
  Interventions: Dietary Supplement: CoQ10; Behavioral: Observational
- HB HIIT +placebo (Placebo Comparator): Participants will receive placebo and home based high intensity interval training for 12 weeks. Exercise will be performed on a non-dialysis day, it will be video-supervised exercise sessions, three days per week for 12 weeks. The three weekly sessions will include: 1 session of 1) body weight high-intensity interval training (bodyweight HIIT), 2) strength training, and 3) walking high-intensity interval training (walking HIIT).
  Interventions: Drug: Placebo; Behavioral: HB-HIIT
- HB HIIT + CoQ10 (Active Comparator): Participants will received CoQ10 1800/day with home based high intensity interval training for 12 weeks. Exercise will be performed on a non-dialysis day, it will be video-supervised exercise sessions, three days per week for 12 weeks The three weekly sessions will include: 1 session of 1) body weight high-intensity interval training (bodyweight HIIT), 2) strength training, and 3) walking high-intensity interval training (walking HIIT).
  Interventions: Dietary Supplement: CoQ10; Behavioral: HB-HIIT

INTERVENTIONS:
Dietary Supplement: CoQ10 — Participants will receive 1800 mg/day for 12 weeks
  Other Names: ubiquinone
  Arms: HB HIIT + CoQ10; Observational+ CoQ10
Drug: Placebo — Participants will receive placebo or CoQ10/day for 12 weeks
  Other Names: inactive substance
  Arms: HB HIIT +placebo; Observational + placebo
Behavioral: HB-HIIT — Participants will be performed on non dialysis days. It will be video supervised exercise sessions with self directed exercises using pre-recorded bodyweight and strength exercise videos.
  Other Names: exercise
  Arms: HB HIIT + CoQ10; HB HIIT +placebo
Behavioral: Observational — Participant regular activities
  Other Names: Normal Routine
  Arms: Observational + placebo; Observational+ CoQ10

SUMMARY:
Frailty and sarcopenia are modifiable risk factors for morbidity and mortality in patients with ESRD. Exercise is the recommended intervention to prevent frailty and sarcopenia, however, many clinical trials have shown limited clinical improvement in muscle mass and physical function. We propose that mitochondrial dysfunction is one of the deterrents to the effectiveness of the exercise. We plan to evaluate the additive effect of HIIT and CoQ10, a mitochondrial-targeted therapy, on mitochondrial function and physical performance. Understanding the interplay among CoQ10, exercise, and mitochondrial function will identify novel mechanisms to improve the efficiency of exercise. This will also serve to prevent frailty, sarcopenia, and muscle dysfunction in patients with ESRD.

DETAILED DESCRIPTION:
Frailty and sarcopenia in patients with end-stage renal disease (ESRD) Patients on maintenance hemodialysis (MHD) experience frailty and sarcopenia. Approximately 73% of patients are diagnosed with frailty at the time of initiation of dialysis. Frailty is a multisystem impairment associated with vulnerability to stressors, and it is characterized by the presence of three of the following criteria: unintentional weight loss, self-reported exhaustion or fatigue, measured muscle weakness, slow walking speed, and low physical activity. The prevalence of frailty increases with age; approximately 7% of individuals older than 65 years of age are diagnosed as frail. Frailty is present at younger ages in patients with ESRD on MHD than in the general population, as many as 44% of patients with ESRD younger than 40 years are frail. Sarcopenia, defined as a reduction in muscle and/or muscle strength, is common in patients on MHD and contributes significantly to the frailty syndrome in this population.6 The loss of muscle power is one of the components of the frailty phenotype, and poor muscle function is recognized as a major cause of frailty.

Muscle mass has been used as a surrogate of muscle function. While the decrease in muscle mass usually correlates with a decrease in muscle strength,11 recent studies have shown that the loss of muscle mass does not fully explain the decrease in muscle function. Likewise, a study in older individuals has shown that the decline in strength is faster than the decline in muscle mass. Furthermore, the maintenance of muscle mass does not necessarily prevent the loss of muscle function, suggesting that the quality of the muscle may play an important role in muscle function. Muscle abnormalities, such as fat infiltration and fibrosis, could explain in part the discrepancy between muscle mass and function. Lack of physical activity is a possible cause of increased intermuscular fat. A study showed that unilateral leg suspension augmented intermuscular fat in thigh muscles. In contrast, aerobic exercise combined with weight loss decreases intermuscular fat. A previous study showed increased intermuscular fat in patients with ESRD compared to controls, a finding we have also observed in our studies. Our preliminary data also showed that intermuscular fat inversely correlates with physical function in patients with ESRD, highlighting the need to find strategies that improve muscle quality and physical function in this population.

Exercise in ESRD Patients with ESRD have reduced muscle mass and strength compared to controls. Resistance exercise is considered the best type of exercise to increase muscle mass and muscle strength. Multiple studies have evaluated the effects of resistance exercise on muscle mass and strength. In most of these studies, resistance exercise failed to elicit an appropriate response compared to the general population. A recent study, using progressive resistance exercise training, showed a comparable increase in muscle mass between healthy controls and patients with ESRD, but it failed to show an improvement in physical function. A single bout of resistance exercise increased muscle protein anabolic effects; however, long-term effects seem to be stalled in patients with ESRD. Many other studies have evaluated the effect of aerobic exercise on peak oxygen consumption (V̇O2peak) in patients with ESRD. These studies showed that on average V̇O2peak increased by 17%, however, this improvement is still less than the predicted age-adjusted V̇O2peak. These data suggest that different exercise strategies need to be tested to examine improvements in physical function.

High-intensity interval training (HIIT) is a particular type of exercise that consists of cycles of brief, high-intensity exercise followed by a recovery period.35 During the period of high intensity, the target is to reach 75% or more of the peak power output. HIIT has been largely unexplored in patients with ESRD. Only one previous pilot study showed that HIIT is feasible and increased peak power output and physical function, but no change in muscle mass.in patients with ESRD on MHD. The benefits of HIIT over other types of exercise regimens (e.g. resistance exercise) reside in its ability to induce mitochondrial biogenesis and improve mitochondrial function. However, it is still unknown if the mitochondrial changes induced by HIIT also occur in patients with ESRD.

Mitochondrial abnormalities in skeletal muscle in patients with ESRD Mitochondria are critical for muscle metabolism and function. We and others have previously shown that mitochondrial abnormalities in skeletal muscle are present in patients with ESRD. These abnormalities include a decreased activity of mitochondrial enzymes, such as citrate synthase and hydroxy acyl-CoA dehydrogenase, and abnormal mitochondrial ultrastructure. We also found that the mitochondrial content is reduced in patients with ESRD, probably due to increased mitophagy and inappropriate mitochondrial biogenesis (generation of new mitochondria). Interestingly, a recent study in a mouse model of CKD showed that reduction in skeletal muscle mitochondrial content would precede the onset of sarcopenia. Recent studies also suggest that mitochondrial dysfunction may play a role in the pathophysiology of sarcopenia. Thus, therapeutic strategies aiming to preserve mitochondrial number and function could be important in preventing the reduction of muscle mass and function in patients with ESRD.

Exercise improves mitochondrial function and induces mitochondrial biogenesis in young and older healthy individuals. On the other hand, mitochondrial dysfunction reduces exercise efficiency and muscle performance. Only three previous studies have evaluated the effect of exercise on mitochondrial biology in patients with CKD. One study showed that exercise prevented the decline in mitochondrial DNA copy number rather than increasing mitochondrial biogenesis. Another study found a numerical but non-significant 15% increase in succinate dehydrogenase (SDH) activity after 20 weeks of endurance training. This change in SDH activity, as mentioned by the authors, is relatively small compared to the increase of 40% or greater in healthy individuals after endurance exercise training. A recent study found that aerobic exercise training increased mitochondrial enzyme activities, but this did not correlate with changes in V̇O2peak. These data suggest that exercise-induced intrinsic mitochondrial changes could be impaired in patients with ESRD on MHD. Changes in mitochondrial dynamics (i.e., fusion and fission of mitochondria) also occur in response to exercise. Mitochondrial fusion leads to enlarged mitochondria and maximizes the oxidative capacity. Mitochondrial fission results in smaller mitochondria and is crucial for the segregation and elimination of damaged mitochondria.68 Previous studies in humans have shown that exercise upregulates both mitochondrial fusion and fission, however, the effects of exercise on mitochondrial dynamics in patients with ESRD remains largely unexplored.

Coenzyme Q10 (CoQ10) as a strategy to restore mitochondrial and muscle function in ESRD The use of mitochondrial-targeted therapies is an obvious approach to improve mitochondrial function and consequently muscle function. CoQ10 (also called ubiquinone) improves mitochondrial function by increasing the coupling of oxidative phosphorylation and oxygen consumption. CoQ10 supplementation has been used in conditions associated with mitochondrial dysfunction, in patients with hypertension, and in statin-induced myopathy. CoQ10 has also been used to improve muscle function. Several studies have explored the effect of CoQ10 supplementation in conjunction with exercise training, showing that CoQ10 increases the anaerobic threshold and peak oxygen consumption. Several other studies found no effect of CoQ10 on exercise capacity, however, these studies were conducted in individuals with normal levels of CoQ10. The effects of CoQ10 have been proven beneficial in individuals with low plasma levels of CoQ10, such as elderly individuals on statin therapy and in patients with heart failure. In the latter group, CoQ10 supplementation reduced mortality and improved functional status, Also, there is an interactive effect of CoQ10 and exercise in patients with heart failure. We and others have observed low levels of plasma CoQ10 in patients with ESRD.24, We also observed an association between CoQ10 redox ratio and mitochondrial function in patients with ESRD (see preliminary data). Our group found that CoQ10 supplementation increases CoQ10 plasma levels and improves the CoQ10 redox ratio in a dose-dependent manner. In a series of studies, our group has also shown that CoQ10 supplementation reduces isofurans and the ratio of isofurans to F2-isoprostanes in patients with ESRD, which are potential markers of mitochondrial dysfunction.

A recent systematic review and meta-analysis have summarized the evidence of CoQ10 supplementation in patients with CKD, not in hemodialysis, showing that CoQ10 may have a metabolic beneficial effects, but recommending more randomized clinical trials (RCTs) to support its use. In patients on MHD, a couple of studies have shown an antioxidant effect of CoQ10 at similar doses that we propose to use in this study. Another study also found that CoQ10 supplementation has a partial effect on oxidative stress in patients on MHD. In contrast, two different studies have shown that CoQ10 does not affect exercise performance, oxidative stress, or diastolic heart function in patients on MHD. It is important to mention that the latter studies use a lower dose (200 mg/day) than the dose we proposed in this study (1800 mg/day). Also, none of the previous studies have evaluated the combination of exercise and CoQ10 supplementation. Therefore, there is a need for rigorous RCTs to define the effect of CoQ10 in patients on MHD Recently it has been shown that knockout mice for mitofusin 2, a protein involved in mitochondrial fusion, have low levels of mitochondrial CoQ10 and abnormal mitochondrial respiration, a phenotype that can be reversed by CoQ10 supplementation.85 Mitofusin 2 may play a role in exporting newly synthesized CoQ10 out of the mitochondria.86, 87 Thus, abnormal mitochondrial dynamics may explain the low levels of CoQ10 in patients with ESRD. All these data suggest that CoQ10 supplementation represents a novel strategy to improve underlying abnormal mitochondrial function and dynamics, as well as enhance the benefits of exercise in patients with ESRD.

Specific Aim 1: Test the hypothesis that CoQ10 enhances the beneficial effect of exercise on mitochondrial function in patients with ESRD on MHD. We hypothesize that the combination of home-based HIIT (HB-HIIT) and CoQ10 will have an additive effect in improving mitochondrial function. We will assess in vivo skeletal muscle mitochondrial function measured by 31P-magnetic resonance spectroscopy (primary outcome) and physical performance measured by the six-minute walk test (secondary outcome).

Specific Aim 2: Test the hypothesis that a combination of exercise training and CoQ10 will improve ex-vivo mitochondrial respiration in patients with ESRD on MHD. For this Aim, muscle biopsies will be performed in patients enrolled in our clinical trial. To evaluate intrinsic changes in mitochondrial function, we will measure mitochondrial respiration (primary outcome) in permeabilized fibers. We will also test the hypothesis that HIIT and CoQ10 combination has an additive effect in increasing mitochondrial content and mitochondrial fusion in patients with ESRD (secondary outcomes). We will also evaluate the transcriptome profiling with RNA sequencing in skeletal muscle to determine if the HIIT and CoQ10 combination upregulates muscle RNA expression of mitochondrial energy metabolism pathways.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 18 to 75 years
* On thrice-weekly chronic hemodialysis for at least 6 months (only applicable for patients with ESRD on maintenance hemodialysis).
* Clinically stable, adequately dialyzed (single-pool Kt/V >1.2) thrice weekly, for at least 3 consecutive months prior to the study (only applicable for patients with ESRD on maintenance hemodialysis)

Exclusion Criteria:

* Body mass index > 35 mg/kg2
* History of functional transplant less than 6 months prior to study
* Use of immunosuppressive drugs within 1 month prior to study
* Active connective tissue disease
* Acute infectious disease within 1 month prior to study
* AIDS (HIV seropositivity is not an exclusion criterion)
* Acute myocardial infarction or cerebrovascular event within 3 months
* Uncontrolled blood pressure
* New or worsening mitral regurgitation murmur
* Hypotension, bradycardia, or tachycardia
* Prolonged ongoing (greater than 20 minutes) angina at rest
* Angina at rest with transient ST changes greater than 0.05 mV on ECG
* Sustained ventricular tachycardia on ECG
* Elevated cardiac enzymes (e.g., troponin Tor I greater than 0.1mg/ml)
* Advanced liver disease, with a modified Child-Turcotte-Pugh score equal or greater than 10.
* Gastrointestinal dysfunction requiring parental nutrition
* Active malignancy excluding basal cell carcinoma of the skin
* Ejection fraction less than 30%
* Pre-dialysis potassium repeatedly higher than 5.5 mmol/L (confirmed on a repeated blood draw)
* Anticipated live donor kidney transplant
* History of poor adherence to hemodialysis or medical regimen
* Inability to provide consent
* Subjects with cardiac pacemaker, artificial heart valve, any metallic implant, permanent tattoo, or any retained foreign metallic bodies.
* Inability to perform exercise
* Contraindication for exercise such as electrolyte abnormalities, uncontrolled arrhythmias, or pulmonary congestion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2027-06-20 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
PCr recovery measured by 31 phosphorus magnetic resonance spectroscopy | 12 weeks
  ERSD 38.7 +/- 5.9 seconds ,with HIIT alone 3.87 sec, with HIIT and CoQ10 11.61.sec

SECONDARY OUTCOMES:
Six minute walk test | 12 weeks
  ESRD 448.1+/-73.7, with exercise alone 8% improvement, with 6MWT and CoQ10 increase by 20%

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Gamboa, MD/PhD, Principal Investigator — VUMC; Talat Ikizler, MD, Principal Investigator — VUMC; Baback Roshanravan, MD/MPH, Principal Investigator — University of California, Davis
Locations (2):
- United States (2):
  - University of California Davis Health, Sacramento, California
  - Vanderbilt University Medical Center-GCRC, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No